CLINICAL TRIAL: NCT03243916
Title: A Prospective Single-arm Study on Targeted and Staged Cyber Knife Combined With Interventional Therapy in the Treatment of Massive Hepatocellular Carcinoma
Brief Title: Targeted and Staged Cyber Knife Combined With Interventional Therapy in the Treatment of MHCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, YuLi, Vice Director of Department of Radiotherappy, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChinaPLAGH-MHCC
Record Dates: First submitted 2017-08-06; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: interventional therapy; TACE; Cyberknife
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combination (Experimental): TACE plus cyber knife
  Interventions: Radiation: TACE plus Cyber knife

INTERVENTIONS:
Radiation: TACE plus Cyber knife — Patients with histologically confirmed MHCC(Massive Hepatocellular Carcinoma) will receive TACE therapy,after 1 or 2 week's recovery from hepatic insufficiency ,the targeted and staged cyber knife will be given

SUMMARY:
Hepatocellular carcinoma is a highly malignant tumor that is progressing rapidly. Hepatic arterial embolization chemotherapy (TACE) is a common method for the treatment of unresectable of hepatocellular carcinoma.But for patients with > 10cm hepatocellular carcinoma, the intervention effect was not satisfied.The cyberknife is a kind of stereotactic radiotherapy which can track the movement of tumor and monitor the position deviation of tumor in real time.This stuy is aimed to observe the efficiency and safety of the combination of TACE and cyberknife in the treatment of massive hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed hepatocellular carcinoma
* No lymph node metastasis or distant metastasis
* Tumor diameter at least 10 cm
* Hepatic lesions are not suitable for surgical resection or the patient refuse to surgical treatment
* Eastern Clinical Oncology Group (ECOG)score is 0， 1or2
* No history of abdominal radiotherapy
* Inoperable and untransplantable,Child-pugh score A or B
* Normal liver volume exceeds 700 cm3

Exclusion Criteria:

* Previous history of abdominal radiotherapy;
* The maximum diameter of tumor is less than 10cm;
* The liver Child is graded C;
* Contraindication for radiotherapy;
* Active gastrointestinal bleeding occurred within 2 weeks before enrollment
* Pregnancy
* Undergoing chemotherapy throughout the past six months
* Diffuse hepatocellular carcinoma
* Main portal vein tumor embolization
* Undergoing other simultaneous treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-08-15 (Estimated); Primary Completion 2019-07-14 (Estimated); Study Completion 2020-07-14 (Estimated)

PRIMARY OUTCOMES:
response rate(RR) | 18 months
  CR(complete response)+PR(partial response)
overall survival(OS) | 26mounth
  Overall survival was defined as the time from enrollment to death from any cause.

SECONDARY OUTCOMES:
adverse event(AE) | 36 month
  Progression Free Survival is defined as the time from enrollment to the date of first documented disease progression or death from any cause
Quality of life (QOL) | 36 month
  A questionnaire with questions referred to simple assessments of physical abilities

CONTACTS AND LOCATIONS:
Overall Officials: Yu Li, MD, Principal Investigator — China PLA hospital
Locations (1):
- Chinese PLA Gereral Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided